CLINICAL TRIAL: NCT05678387
Title: Gut Microbiota in Adults With Chronic Widespread Pain: a Pilot Case-control Study
Brief Title: Gut Microbiota in Adults With Chronic Widespread Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Regina Wing Shan Sit, Prof. Regina Wing Shan SIT, Chinese University of Hong Kong
Other Study IDs: 2022.469
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Chronic Widespread Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The de-identified stool sample specimens left from this study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants: Participants without chronic pain and depression
- Chronic Widespread Pain participants: Participants with Chronic Widespread Pain

SUMMARY:
We aim to identify the gut microbiome composition in adults with CWP. We will collect the stool sample of 120 healthy individuals and 120 Chronic Widespread Pain patients. We hypothesize that the intestinal microbiota is altered in CWP compared to healthy subjects without CWP.

DETAILED DESCRIPTION:
We aim to identify the variations in gut microbiota composition in Hong Kong adults with CWP. We hypothesize that the intestinal microbiota is altered in CWP compared to healthy control. The design of the study is a pilot case-control study with adults with CWP (n=120) and healthy adults without any chronic pain (n=120). Participants will be recruited in 8 general-outpatient clinics in the New Territories East region of Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with Chronic Widespread pain

   Participants will be asked, "In the past 3 months, have you had pain in your muscles, bones and joints lasting at least 1 week?", as a screening question for CWP. To meet the criteria for CWP, subjects have to report musculoskeletal pain in at least 4 of 5 body regions and in at least 3 or more body quadrants (as defined by upper-lower/left-right side of the body) and axial skeleton (neck, back, chest, and abdomen), with pain duration of more than 3 months. A Widespread Pain Index (WPI) will be generated based on the number of pain sites. Subgroup of patients with fibromyalgia will be identified according to The American College of Rheumatology 2016 when subjects WPI of ≥ 7 and a symptom severity scale (SSS) score of ≥ 5 or a WPI between 4 and 6 and an SSS score of ≥ 9.
2. Healthy Participants

Healthy participants will be those without chronic pain and depression. A screening question 'In the past 3 months, have you had pain in your muscles, bones and joints lasting at least 1 week?' will be asked to determine whether participant has chronic pain. Depression status will be determined by the questionnaire "Patient Health Questionnaire-9"

Exclusion Criteria:

* Participants with major chronic illnesses, such as malignancy, active inflammatory diseases, autoimmune diseases and metabolic diseases such as diabetes mellitus and thyroid diseases etc.; use of antibiotics, probiotics or prebiotics in the preceding 2 months, any acute illness in the preceding month, change in regularly taken medication in the preceding month, and substantial dietary alterations in the preceding month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited in 8 general-outpatient clinics in the New Territories East region of Hong Kong. Healthy participants with matching age and sex will be recruited from the general public.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome composition | week 1
  The gut microbiome composition of participants with CWP, as compared with healthy participants

OTHER OUTCOMES:
Depressive status | At baseline, study week 0
  The depressive status of participants will be assessed by the Patient Health Questionnaire (PHQ-9), a 9-item self-reported measures to diagnose and assess the severity of depression.
Dietary intake | At study week 1
  Dietary intake will be assessed by the Hong Kong Diet Score (HKDS), a 9-item diet screener, based on Mediterranean Diet Score (MDS) cutoff values and Hong Kong Chinese food consumption reported by the government.
Bowel habit | At study week 1
  Bowel habit will be assessed by the Bristol Stool Scale (BSS), a validated measure of intestinal transit that categorizes stool into 7 types from type 1 (hard lumps) to type 7 (watery diarrhea)
Physical activity level | At study week 1
  Physical activity will be assessed by the Chinese version of International Physical Activity Questionnaire (IPAQ) short form.
Use of Chronic medications | At baseline, study week 0
  The use of chronic medications will be enquired from participants and further confirmed with hospital electronic system.
Sociodemographic data | At baseline, study week 0
  Sociodemographic information such as age and sex, comorbid diseases, lifestyle habits (smoking and drinking status)
BMI | At baseline, study week 0

CONTACTS AND LOCATIONS:
Overall Officials: Regina Wing Shan Sit, Principal Investigator — Jockey Club School of Public Health and Primary Care, Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Shatin, Hong Kong